CLINICAL TRIAL: NCT03489434
Title: Technology-Based Prevention for Adolescents in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Responsible Party: Principal Investigator, Amanda Gilmore, Assistant Professor, Georgia State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H21524
Record Dates: First submitted 2018-03-29; First posted 2018-04-05 (Actual); Results first posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Substance Use
Keywords: adolescents; primary care; sexual assault; substance use; sexual risk behavior
MeSH Terms: conditions — Substance-Related Disorders | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participant and Investigator are blinded to condition
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Preliminary prevention program component content is based on evidence-based prevention programs and will integrate prevention content for substance use, sexual assault, and sexual risk behaviors.
  Interventions: Behavioral: Intervention
- Control (No Intervention): Assessment only control.

INTERVENTIONS:
Behavioral: Intervention — Preliminary prevention program component content is based on evidence-based prevention programs and will integrate prevention content for substance use, sexual assault, and sexual risk behaviors.
  Arms: Intervention Group

SUMMARY:
Adolescent substance use, sexual assault, and sexual risk behaviors pose a great public health concern, and subsequently there is also a great need to prevent these behaviors and experiences. This project involves the adaptation and integration of evidence-based prevention content aimed at preventing and reducing substance use, sexual assault, and sexual risk behaviors. This project uses innovative technology within primary care visits to conduct a feasibility trial of an integrated prevention program.

DETAILED DESCRIPTION:
Pilot feasibility trial in preparation for RCT. Adolescents aged 14-18 will be recruited for screening from community-based primary care clinics to ensure ease of dissemination and representation of community-based primary care settings. The primary goal is to develop feasibility to apply for an R01 to conduct an RCT. Power analyses indicate that 280 participants would be needed for an RCT after accounting for attrition. Given that the RCT would be conducted over a 3-year period, a recruitment rate of 8 adolescents per month would indicate feasibility for a larger RCT.

ELIGIBILITY:
Inclusion Criteria:

* Aged 14-18
* Recent visit to primary care doctor

Exclusion Criteria:

* Inability to comprehend English independently due to disability or language

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 123 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda K Gilmore, PhD, Principal Investigator — Georgia State University
Locations (1):
- Georgia State University, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Gilmore AK, Fortson K, Mullican KN, Garcia-Ramirez G, Hutchins A, Bartlett AM, Gooding HC, Wallis E, Levy S, Ruggiero KJ, Kaysen D, Danielson CK, Platner R, Hartman A, Self-Brown S. An eHealth Prevention Program for Substance Use, Sexual Assault, and Sexual Risk Behaviors for Adolescents in Primary Care: Pilot Feasibility Randomized Controlled Trial of Teen Well Check. JMIR Form Res. 2023 Nov 2;7:e50833. doi: 10.2196/50833. PMID 37917146

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Group | Control
Started | 61 | 62
Completed | 55 | 40
Not Completed | 6 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control | Total
Number analyzed (Participants) | 61 | 62 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.62 (1.39) | 15.63 (1.24) | 15.63 (1.31)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Boy | 31 | 27 | 58
  Girl | 28 | 34 | 62
  Nonbinary | 2 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 1
  Black or African American | 59 | 58 | 117
  White | 2 | 1 | 3
  Not listed or prefer not to answer | 0 | 2 | 2
  Hispanic or Latine | 1 | 4 | 5
  Not Hispanic or Latine | 46 | 50 | 96
Region of Enrollment [Number; unit: participants]
  United States | 61 | 62 | 123
Substance Use Risk [Count of Participants; unit: Participants]
  Alcohol | 8 | 8 | 16
  Cannabis | 8 | 12 | 20
  Tobacco or vaping | 5 | 5 | 10
  Prescription drug misuse | 8 | 8 | 16
  Illegal drugs | 2 | 1 | 3
Ever engaged in sex [Count of Participants; unit: Participants] | 14 | 13 | 27
Substance use before sex in past 90 days [Count of Participants; unit: Participants] | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Enrollment and Recruitment Rate
Description: Feasibility of enrollment recruitment was assessed by the proportion of anticipated participants enrolled in the study
Time Frame: within 2 year recruitment period
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control
Number analyzed (Participants) | 61 | 62
Participants | 61 | 62

2. Primary Outcome: Retention Rate: Number of Participants Who Completed at Least 1 Follow-Up Study
Description: Feasibility of retention was assessed by the proportion of participants retained in the study
Time Frame: within 6 months of baseline participation
Measure: Count of Participants; unit: Participants
Groups:
- Intervention: Retention for the intervention condition was calculated using the number of participants who completed at least one follow-up study.
- Control: Retention for the control condition was calculated using the number of participants who completed at least one follow-up study.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 61 | 62
Participants | 50 | 54

ADVERSE EVENTS:
Time Frame: Adverse events were monitored over the 6-month data collection period.
Arm/Group | Intervention Group | Control
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/62
Other Adverse Events (participants affected / at risk) | 0/61 | 0/62

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/34/NCT03489434/Prot_SAP_001.pdf
  • Informed Consent Form (2021-09-16): https://cdn.clinicaltrials.gov/large-docs/34/NCT03489434/ICF_002.pdf